CLINICAL TRIAL: NCT00832247
Title: Phase 1 Study of Autologous Bone Marrow Mononuclear Cells Infusion in Peripheral Vein in Liver Cirrhosis Due to Hepatitis C Virus
Brief Title: Autologous Bone Marrow Mononuclear Cells in Liver Cirrhosis
Acronym: CELTHEP-02
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado do Rio de Janeiro (FAPERJ) (Unknown); Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government); Financiadora de Estudos e Projetos (Other); Oswaldo Cruz Foundation (Other); University of Edinburgh (Other)
Responsible Party: Guilherme Ferreira da Motta Rezende, Federal UNiversity of Rio de Janeiro
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CELTHEP-02
Record Dates: First submitted 2009-01-29; First posted 2009-01-30 (Estimated); Last update posted 2009-01-30 (Estimated); Status verified 2009-01

CONDITIONS: Liver Cirrhosis Due to Virus C Chronic Hepatitis
Keywords: Hepatitis C; Cirrhosis; Stem cell
MeSH Terms: conditions — Hepatitis C; Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Genetic: Autologous bone marrow mononuclear cells infusion — At least 100.000.000 autologous BMMC will be infused in a peripheral vein once suspended in albumine during 10 minutes

SUMMARY:
This is a phase I clinical study to evaluate feasibility, safety and kinetics of cellular therapy with autologous bone marrow-derived mononuclear cells (BMMC) in patients with liver cirrhosis due to virus C hepatitis. Another aim is to study liver tissue changes induced by the BMMC presence. All the patients have moderate liver disfunction and will be submitted to a liver biopsy before BMMC injection. The cells will be labeled with 99mTc and infused through a peripheral vein. Scintigraphy will be performed 24 hours after infusion.

Patients will be submitted to frequent clinical, laboratorial and image evaluation during a one-year follow-up. A second liver biopsy will be done in the 3rd month after infusion to check histological, cellular and molecular evolutive changes.

ELIGIBILITY:
Inclusion Criteria:

* Chronic virus C hepatitis
* Liver cirrhosis
* Moderate liver disfunction

Exclusion Criteria:

* Malignant disease
* Pregnancy
* Significant comorbidity
* Portal vein thrombosis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2009-01; Primary Completion 2010-04 (Estimated); Study Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
Liver function worsening | One year

SECONDARY OUTCOMES:
Liver related mortality | One year
Hepatocellular carcinoma development accessed by ultrasound and CT scan | One year
BMMC kinetics accessed by total body scintigraphy | 24 hours
Liver tissue changes evaluated by histopathology analysis and molecular biology | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Guilherme FM Rezende, MD PhD, Principal Investigator — Universidade Federal do Rio de Janeiro
Locations (1):
- Hospital Universitário Clementino Fraga Filho, Rio de Janeiro, Rio de Janeiro, Brazil